CLINICAL TRIAL: NCT00197639
Title: A Pharmacokinetic Study to Assess the Inter-patient Variability of Indinavir Drug Levels When Boosted With Ritonavir in Thai Patients on Highly Active Antiretroviral Therapy
Brief Title: Pharmacokinetic Study of Indinavir Drug Levels When Boosted With Ritonavir in Thailand
Status: Completed | Type: Observational
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Other Study IDs: HSC 10913; R01HD042964 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2010-11-15 (Estimated); Status verified 2010-11

CONDITIONS: HIV Infection
Keywords: indinavir, HIV, ritonavir, pharmacokinetics, Thailand
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ritonavir-boosted indinavir

SUMMARY:
This study looks at the ways indinavir drug levels, when boosted with ritonavir, may vary from patient to patient. The study population are HIV+ Thai individuals.

DETAILED DESCRIPTION:
This study will assess the inter-individual variability of indinavir drug levels, boosted with ritonavir, in Thai patients. Data will be collected in patients participating in the randomized study, "Monitoring Highly Active Antiretroviral Therapy (HAART) in HIV-infected patients in Thailand (PHPT-3)" (HSC 10668). The first 20 patents in PHPT-3 will have steady-state pharmacokinetic sparse sampling performed at pre-dose, and 1, 2.5, 4 and 12 hours after drug intake 1 and 2 months after initiating IDV/r 400/100 mg, twice daily. IDV/r plasma concentrations will be determined by high performance liquid chromatography. This spare PK data will be pooled with indinavir concentration data collected within an intensive pharmacokinetic studies of IDV/r [Cressey TR, et al 2005, JAC, 55, p1041-44]. Population means and variances of indinavir and ritonavir pharmacokinetic parameters were estimated using non-linear mixed effects regression models (NONMEM Version VI). The validity of the final model was evaluated using a visual predictive check (VPC) and bootstrap re-sampling techniques.

ELIGIBILITY:
Inclusion Criteria:

* Subjects enrolled in the parent study, "Monitoring HAART Therapy in HIV-Infected Patients in Thailand (PHPT-3)" and agreeing to additional blood sampling and tests.

Exclusion Criteria:

* Current active substance or alcohol abuse
* Active opportunistic infection
* Chronic malabsorption or diarrhea
* Other clinically significant disease
* Certain lab values (e.g. hemoglobin < 8.0 mg/dL)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: HIV-infected Thai adults
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2006-09; Primary Completion 2009-05 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Lallemant, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (4):
- Thailand (4):
  - Prapokklao Hospital, Muang, Changwat Chanthaburi
  - Chonburi Hospital, Muang, Changwat Chon Buri
  - Phayao Provincial Hospital, Muang, Changwat Phayao
  - Nakornping Hospital, Mae Rim, Chiang Mai

REFERENCES:
- [Background] Cressey TR, Leenasirimakul P, Jourdain G, Tod M, Sukrakanchana PO, Kunkeaw S, Puttimit C, Lallemant M. Low-doses of indinavir boosted with ritonavir in HIV-infected Thai patients: pharmacokinetics, efficacy and tolerability. J Antimicrob Chemother. 2005 Jun;55(6):1041-4. doi: 10.1093/jac/dki143. Epub 2005 May 9. PMID 15883177